CLINICAL TRIAL: NCT00625066
Title: Tennessee Colorectal Polyp Study
Brief Title: Biological, Genetic, and Lifestyle Risk Factors for Developing Colorectal Adenomas or Polyps in Participants Undergoing Colonoscopy
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wei Zheng, Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: CDR0000583154; P30CA068485 (NIH); VU-VICC-GI-0294; VU-VICC-020603; VU-VICC-020531
Record Dates: First submitted 2008-02-27; First posted 2008-02-28 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Precancerous Condition
Keywords: precancerous condition; colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Colonic Neoplasms; Rectal Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: biologic sample preservation procedure
Other: cytology specimen collection procedure
Other: medical chart review
Other: questionnaire administration
Other: survey administration
Procedure: biopsy
Procedure: evaluation of cancer risk factors
Procedure: screening colonoscopy

SUMMARY:
RATIONALE: Collecting and storing samples of tissue, blood, and other body fluids to test in the laboratory and gathering information about health and lifestyle from participants may help doctors learn more about cancer risk factors.

PURPOSE: This clinical trial is looking at biological, genetic, and lifestyle risk factors for developing colorectal adenomas or polyps in participants undergoing colonoscopy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To recruit 7,000 participants who are planning to undergo colonoscopy.
* To collect questionnaires and medical records from these participants.
* To collect biological samples, including urine, blood, buccal cells and/or saliva, rectal tissue, and colorectal polyps from these participants.
* To evaluate risk factors and other differences between participants found to have polyps and those who do not have polyps.

OUTLINE: Participants undergo screening colonoscopy and removal of any polyps.

Within 1 month of colonoscopy, participants undergo a 30-minute telephone interview and/or complete a mail survey to provide information on lifestyle and medical history that may be related to colorectal polyp risk. Participants who undergo removal of polyps during their colonoscopy also complete a 20-minute survey at their 3-year follow-up colonoscopy. Participants' medical records may also be reviewed.

Blood samples are collected at the time of colonoscopy. Some participants may also provide blood samples 1-2 weeks prior to colonoscopy. Tissue from the bisected portions of colorectal polyps > 5 mm in size that are removed during colonoscopy is also obtained. Some participants may also undergo normal colorectal tissue sample and saliva sample collection at the time of colonoscopy and urine sample collection 2 days prior to, during, and/or 8 weeks after colonoscopy.

Tissue samples may be stored for future genetic studies to evaluate genetic factors that may cause or be related to colon polyps or colorectal cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Scheduled to undergo colonoscopy at the Vanderbilt University Medical Center or the Tennessee Valley Veterans Administration Medical Center
* No prior genetic colorectal cancer syndromes or colorectal adenoma

PATIENT CHARACTERISTICS:

* Must have a permanent residence and a telephone number
* Able to speak and understand English
* No prior inflammatory bowel disease
* No prior cancer other than nonmelanoma skin cancer
* Not a current resident in a correctional facility
* No other rare exclusion that would prevent the collection of study data (e.g., extensive memory loss for past exposures), impair ability to provide informed consent, or make the participant an atypical colonoscopy patient (e.g., colonoscopy for organ transplant evaluation)
* No prior extensive knowledge or contact with the investigation/protocol/hypotheses (the study collaborator or reviewer)

PRIOR CONCURRENT THERAPY:

* No prior partial or complete colon resection
* No concurrent participation in a clinical trial involving the prevention of colon polyps

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants who are planning to undergo colonoscopy
Sampling Method: Probability Sample
Enrollment: 8108 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Recruitment of 7,000 participants who are planning to undergo colonoscopy
Collection of questionnaires and medical records
Collection of biological samples, including urine, blood, buccal cells and/or saliva, rectal tissue, and colorectal polyps
Evaluation of risk factors and other differences between participants found to have polyps and those who do not have polyps

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zheng, MD, PhD, MPH, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Murff HJ, Shrubsole MJ, Cai Q, Smalley WE, Dai Q, Milne GL, Ness RM, Zheng W. Dietary intake of PUFAs and colorectal polyp risk. Am J Clin Nutr. 2012 Mar;95(3):703-12. doi: 10.3945/ajcn.111.024000. Epub 2012 Jan 25. PMID 22277551